CLINICAL TRIAL: NCT05417672
Title: Assessment of Relationship Between Preoperative Nutritional Status and Perioperative/Postoperative Conditions in Patients With Lung Cancer Scheduled for Lobectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turkish Society of Anesthesiology and Reanimation (Other)
Responsible Party: Sponsor
Other Study IDs: LungCancerMalnutrition
Record Dates: First submitted 2022-06-02; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Lung Cancer; Malnutrition; Nutritional Deficiency
MeSH Terms: conditions — Lung Neoplasms; Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung cancer scheduled lobectomy
  Interventions: Diagnostic Test: Nutritional Risk Screening-2002; Diagnostic Test: Nutritional Risk Index; Diagnostic Test: Mini Nutritional Assessment; Diagnostic Test: Glasgow Prognostic Score; Diagnostic Test: Prognostic Nutritional Index; Diagnostic Test: Anthropometric measurements; Device: Handgrip strength test

INTERVENTIONS:
Diagnostic Test: Nutritional Risk Screening-2002 — Nutritional Risk Screening-2002
Diagnostic Test: Nutritional Risk Index — Nutritional Risk Index
Diagnostic Test: Mini Nutritional Assessment — Mini Nutritional Assessment
Diagnostic Test: Glasgow Prognostic Score — Glasgow Prognostic Score
Diagnostic Test: Prognostic Nutritional Index — Prognostic Nutritional Index
Diagnostic Test: Anthropometric measurements — middle arm circumference
Device: Handgrip strength test — Handgrip strength test

SUMMARY:
Malnutrition is common in patients with lung cancer. In patients with malnutrition risk, the risk of complications is high both in the perioperative, early and late postoperative periods. Malnutrition is an independent risk factor for length of hospital stay and cost in these patients. Patients with lung cancer may have many morbidities in postoperative period, especially problems with wound healing. Therefore, assessment of the nutritional status of patients with lung cancer should begin at the diagnosis stage.

DETAILED DESCRIPTION:
In patients with lung cancer scheduled for lobectomy, anthropometric measurements will be measured and the results of laboratory tests(albumin, prealbumin, creatinine, total lymphocyte count, C reactive protein), Nutritional Risk Screening-2002, Nutritional Risk Index, Mini Nutritional Assessment, Glasgow Prognostic Score, Prognostic Nutritional Index and neoadjuvant chemotherapy or not will be recorded in 72 hours before surgery. In addition, demographic information of the patients (name, surname, identification number, age, comorbidity, American Society of Anesthesiologists score) will be recorded. After the information is given to the patients, their written and verbal consent will be obtained.

In the operating room, routine monitoring (electrocardiography, invasive blood pressure measurement, arterial blood gas monitoring, peripheral oxygen saturation, end-tidal carbon dioxide measurement by capnography) will be applied to the patients in accordance with the standard protocol for elective lobectomy surgery.

Hemodynamic changes (eg. dysrhythmia, hypotension, hypertension, hemorrhage), metabolic status (pH, bicarbonate, base excess), lactate, glucose level in blood gas evaluation and intraoperative complications will be recorded during the intraoperative period.

In the postoperative period, length of stay in the intensive care unit, length of hospital stay, early complications (eg. dysrhythmia, acute coronary syndrome, sepsis, mediastinitis, pneumonia, surgical site infection, prolonged air leak), time to start oral intake and transition to adequate oral intake will be recorded in the one-month postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of lung cancer
* Lung lobectomy operation will be performed
* 18 years and older patients
* Having an American Society of Anesthesiologists score of 1, 2, 3
* Having approved and signed the informed consent form

Exclusion Criteria:

* Patients who underwent lobectomy with a diagnosis other than lung cancer
* Patients younger than 18 years
* Patients with an American Society of Anesthesiologists score of 4 and above
* Patients who did not accept informed consent
* Patients who refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years and older patients who underwent lobectomy with a diagnosis lung cancer
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-06-08 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | a month after the surgery
  dysrhythmia, acute coronary syndrome, sepsis, mediastinitis, pneumonia, surgical site infection, prolonged air leak
Length of stay in the intensive care unit | up to 30 days
  Length of stay in the intensive care unit
Length of hospital stay | up to 30 days
  Length of hospital stay
Intraoperative hemodynamic complications | during the procedure
  dysrhythmia, hypotension, hypertension, hemorrhage

SECONDARY OUTCOMES:
Oral intake | up to 30 days
  time to start oral intake and transition to adequate oral intake
pH | during the procedure
  pH in arterial blood gas evaluation
bicarbonate | during the procedure
  bicarbonate level in arterial blood gas evaluation
base excess | during the procedure
  base excess in arterial blood gas evaluation
lactate | during the procedure
  lactate level in arterial blood gas evaluation
glucose | during the procedure
  glucose level in arterial blood gas evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludağ Üniversitesi Tıp Fakültesi, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cederholm T, Barazzoni R, Austin P, Ballmer P, Biolo G, Bischoff SC, Compher C, Correia I, Higashiguchi T, Holst M, Jensen GL, Malone A, Muscaritoli M, Nyulasi I, Pirlich M, Rothenberg E, Schindler K, Schneider SM, de van der Schueren MA, Sieber C, Valentini L, Yu JC, Van Gossum A, Singer P. ESPEN guidelines on definitions and terminology of clinical nutrition. Clin Nutr. 2017 Feb;36(1):49-64. doi: 10.1016/j.clnu.2016.09.004. Epub 2016 Sep 14. PMID 27642056
- [Background] McKenna NP, Bews KA, Al-Refaie WB, Colibaseanu DT, Pemberton JH, Cima RR, Habermann EB. Assessing Malnutrition Before Major Oncologic Surgery: One Size Does Not Fit All. J Am Coll Surg. 2020 Apr;230(4):451-460. doi: 10.1016/j.jamcollsurg.2019.12.034. Epub 2020 Feb 26. PMID 32113029
- [Background] Detsky AS, McLaughlin JR, Baker JP, Johnston N, Whittaker S, Mendelson RA, Jeejeebhoy KN. What is subjective global assessment of nutritional status? JPEN J Parenter Enteral Nutr. 1987 Jan-Feb;11(1):8-13. doi: 10.1177/014860718701100108. PMID 3820522
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Background] Vellas B, Guigoz Y, Garry PJ, Nourhashemi F, Bennahum D, Lauque S, Albarede JL. The Mini Nutritional Assessment (MNA) and its use in grading the nutritional state of elderly patients. Nutrition. 1999 Feb;15(2):116-22. doi: 10.1016/s0899-9007(98)00171-3. PMID 9990575
- [Background] Neelemaat F, Kruizenga HM, de Vet HC, Seidell JC, Butterman M, van Bokhorst-de van der Schueren MA. Screening malnutrition in hospital outpatients. Can the SNAQ malnutrition screening tool also be applied to this population? Clin Nutr. 2008 Jun;27(3):439-46. doi: 10.1016/j.clnu.2008.02.002. Epub 2008 Apr 18. PMID 18395946